CLINICAL TRIAL: NCT06520592
Title: Using Augmented Reality to Establish and Evaluate the Effectiveness of a Set of Continuous Positive Airway Pressure Care Management Protocol for Obstructive Sleep Apnea Patients
Brief Title: The Effectiveness of Augmented Reality to Enhance CPAP Therapy in OSA Patients
Acronym: CPAP OSA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chen, Yen-Chin, Associate Professor, National Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: A-ER-111-531; 112-2628-B-110 -006 -MY3 (Other Grant/Funding Number: National Science and Technology Council)
Record Dates: First submitted 2024-07-20; First posted 2024-07-25 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2024-08

CONDITIONS: Aherence; Physical Symptoms; Mental Health; Quality of Life
Keywords: Augmented Reality (AR); continuous positive airway pressure (CPAP); Adherence; Symptoms change
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: For the interventional group, they will utilize AR-guided CPAP therapy to ensure a proper fit of the CPAP device mask and successful adherence to the CPAP therapy. For the standard of care group, they will receive the standard of care.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participnants will be randomly assigned to experimental or control groups by using block randomized method. In the study, we will use independent staff members who are not involved in outcome assessment to handle administrative tasks related to group assignments. In order to mask outcomes assessors, we will ensure that all documents and data sets used by the outcome assessors do not contain any information that could reveal group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With AR guided CPAP therapy (Experimental): OSA patientns were assigned to experimental group, they will be received AR guided CPAP therapy
  Interventions: Behavioral: With AR guided CPAP therapy
- Standard of care (No Intervention): OSA patientns were assigned to stand of care group, they will be not received AR guided CPAP therapy

INTERVENTIONS:
Behavioral: With AR guided CPAP therapy — Participants will received AR training course to utilize the AR guided CPAP therapy
  Arms: With AR guided CPAP therapy

SUMMARY:
The goal of this clinical trial is to exam if artificial reality works to improve continuous positive airway pressure (CPAP) adherence in obstructive sleep apnea (OSA) patients. It will also learn about the feasibility of AR guided CPAP therapy. The main questions it aims to answer are:

Does AR guided CPAP therapy increase the adherence of CPAP therapy among OSA patients? What barriers do participants have when using AR guided CPAP therapy? Researchers will compare AR guided CPAP therapy to a control (standard of care) to see if AR guided CPAP therapy works to enhance the adherence of CPAP therapy.

Participants will:

1. Take AR guided CPAP therapy or standard of care every day for 6 months
2. Visit the clinic on baseline (t0), receiving CPAP therapy at the 1st month (t1), for checkups and tests, receiving CPAP therapy at the 3rd month (t2), receiving CPAP therapy at the 6th month (t3).
3. Response their symptoms on each following time.

DETAILED DESCRIPTION:
Participants will randomly assign to two group, for experimental group will be received AR guided CPAP therapy. In the control group will be received standard of care.

ELIGIBILITY:
Inclusion Criteria:

* (1) Diagnosed with moderate to severe obstructive sleep apnea (AHI≥15) through polysomnography (PSG).
* (2) Age is equal to or greater than 20 years old or equal.

Exclusion Criteria:

* (1) individuals who have previously used positive pressure ventilators for treatment,
* (2) those diagnosed with central sleep apnea,
* (3) those with uncontrolled acute mental illness,
* (4) terminally ill patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The adherence of CPAP therapy | From enrollment to the end of treatment at 6 months
  Adherence refers to the patient's adherence to CPAP therapy, which means using CPAP for more than 70% of the total sleep time during the night, with a minimum duration of 4 hours. The calculation method involves dividing the number of days with CPAP use exceeding 4 hours by the total number of days and multiplying by 100 to obtain the average percentage of CPAP usage.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rotenberg BW, Murariu D, Pang KP. Trends in CPAP adherence over twenty years of data collection: a flattened curve. J Otolaryngol Head Neck Surg. 2016 Aug 19;45(1):43. doi: 10.1186/s40463-016-0156-0. PMID 27542595
- [Background] Bakker JP, Weaver TE, Parthasarathy S, Aloia MS. Adherence to CPAP: What Should We Be Aiming For, and How Can We Get There? Chest. 2019 Jun;155(6):1272-1287. doi: 10.1016/j.chest.2019.01.012. Epub 2019 Jan 23. PMID 30684472
- [Background] Wiederhold BK. How Virtual Reality Is Changing the Reality of Aging. Cyberpsychol Behav Soc Netw. 2020 Mar;23(3):141-142. doi: 10.1089/cyber.2020.29176.bkw. No abstract available. PMID 32150700
- [Derived] Chen MC, Chen YC, Lin CY. Enhancing Adherence to Continuous Positive Airway Pressure Therapy in Patients With Obstructive Sleep Apnea Using Augmented Reality: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 May 6;14:e69757. doi: 10.2196/69757. PMID 40327384